CLINICAL TRIAL: NCT02680886
Title: Post-Marketing Clinical Follow-up (PMCF) Study for Skin Closure to Evaluate the Safety and Efficacy of Novosyn® Quick Suture Material. A Multicenter, International, Prospective, Observational Study
Brief Title: PMCF-study Using Novosyn® Quick Suture Material for Skin Closure
Acronym: SKINNOQ
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1505
Record Dates: First submitted 2016-02-05; First posted 2016-02-12 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-01

CONDITIONS: Skin Closure
Keywords: Rapid Absorbable Suture Material; Children / Adults; Novosyn Quick

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novosyn® Quick: Skin closure using rapid absorbable suture material
  Interventions: Device: Novosyn® Quick

INTERVENTIONS:
Device: Novosyn® Quick — Skin closure

SUMMARY:
The aim of this study is to show that the performance of Novosyn® Quick suture material is comparable with other suture material used for skin closure. In order to show that, various safety and efficacy parameters have been selected. The outcome regarding these parameters will be evaluated by a quantitative summary of the available clinical data from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adult patients undergoing skin closure
* Small linear minimally contaminated incision / lacerations on the trunk or extremities
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Facial lacerations or incisions
* Visible dirt in the wounds
* Nonlinear shape
* Patients taking medical consumption that might affect wound healing

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children and adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Wound infection | 3 months
  Wound infection (Surgical site infection, SSI) is defined according to the definition of the US Centres for Disease Control and Prevention (CDC).
Incidence of wound dehiscence | 3 months postoperatively
  A dehiscence of the skin which needs surgical treatment with re-closure
Incidence of Tissue reaction / Inflammation | 3 months postoperatively
Incidence of Suture removal | 3 months postoperatively
  Suture removal due to insufficient absorption
Incidence of Re-suturing | 3 months post-operatively
  Re-Suturing due to dehiscence
Cosmetic result | 3 months post-operatively
  Cosmetic result after surgery using the Patient and Observer Scar Assessment Scale (POSAS). Cosmetic result and the scar will be evaluated by the patient and the physician. Patient will rate the cosmetic outcome using the patient component of the Patient and Observer Scar Assessment Scale (POSAS). The physician will use the Observer component of the POSAS to assess the cosmetic outcome.
  Documentation of the scar will be performed 3 months postoperatively using photographs.
  Overall patient and observer satisfaction with the scar after 3 months postoperatively (POSAS).
Assessment of the handling of the suture material | intraoperatively
  Assessment of the handling of the suture material intra-operatively using a questionnaire including different dimensions (knot security, tensile strength, knot run down, tissue drag etc.) with 5 evaluations levels (excellent, very good, good, satisfied, poor).

CONTACTS AND LOCATIONS:
Locations (2):
- Hospital Saint Louis, La Rochelle, France
- Klinikum der Johann-Wolfgang-Goethe Universität, Department for Pediatric Surgery and Pediatric Urology, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gfroerer S, Baumann P, Schwalbach AK, Smirnoff A. Prospective international multicenter observational study of Novosyn(R) Quick for skin closures in adults and children (SKINNOQ). BMC Surg. 2019 May 2;19(1):47. doi: 10.1186/s12893-019-0506-8. PMID 31046730